CLINICAL TRIAL: NCT01690819
Title: Protective Ventilatory Strategy in Severe Acute Brain Injury: Randomized Multi-center Controlled Trial
Brief Title: Protective Ventilatory Strategy in Severe Acute Brain Injury
Acronym: PROLABI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Luciana Mascia, MD, PhD, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROLABI
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Injuries, Acute Brain
Keywords: Acute Respiratory Distress Syndrome; Acute Brain Injury
MeSH Terms: conditions — Brain Injuries; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Ventilatory Strategy (Active Comparator): Conventional Ventilatory Strategy
  Interventions: Procedure: Conventional Ventilatory Strategy
- Protective Ventilatory Strategy (Experimental): Protective ventilatory strategy
  Interventions: Procedure: Protective Ventilatory Strategy

INTERVENTIONS:
Procedure: Conventional Ventilatory Strategy — The conventional strategy will be the standard of care with a lower limit of tidal volume equal to 8 ml/Kg of predicted body weight and with a PEEP of 4 cmH2O
  Arms: Conventional Ventilatory Strategy
Procedure: Protective Ventilatory Strategy — The protective strategy will consist of a tidal volume of 6 ml/Kg of predicted body weight, with a PEEP of 8 cmH2O
  Arms: Protective Ventilatory Strategy

SUMMARY:
Acute respiratory distress syndrome (ARDS) occurs in almost 20% of patients with severe acute brain injury and is associated with increased morbidity and mortality. A massive increase in sympathetic activity and an increased production of proinflammatory cytokines released into the systemic circulation are the most important recognized mechanisms. Altered blood brain barrier after injury causes spillover of inflammatory mediators from the brain into the systemic circulation leading to peripheral organs damage. The adrenergic surge induces an increase in vascular hydrostatic pressure and lung capillary permeability, causing an alteration of alveolar capillary barrier with fluid accumulation, resulting in ARDS.

The main goal of mechanical ventilation after acute brain injury are the maintenance of optimal oxygenation, and a tight control of carbon dioxide tension, although ventilatory settings to be used to obtain these targets, while avoiding secondary insults to the brain, are not clearly identified.

Protective ventilatory strategy has been positively evaluated first in patients with ARDS, and then in those undergoing cardiopulmonary bypass or lung resection surgery, or in brain death organ donors, but data on the effect of protective mechanical ventilation on patients with acute brain injury are still lacking even if this is a population with recognized risk factors for ARDS.

Therefore, the primary aim of this multi-center, prospective, randomized, controlled trial is to investigate whether a protective ventilatory strategy, in the early phase after severe acute brain injury, is associated with a lower incidence of ARDS, avoiding any further damage to the brain. Secondary aim is to evaluate if a protective ventilatory strategy is associated with reduced duration of mechanical ventilation, incidence of organ failure, intensive care unit length of stay, and lower concentrations of plasma inflammatory cytokines, without adversely affect in neurological outcome.

DETAILED DESCRIPTION:
BACKGROUND Acute respiratory distress syndrome (ARDS) is described as the most common non-neurologic organ dysfunction occurring in the early phase after severe acute brain injury, with a reported incidence of 10-15% and increased morbidity and mortality.

A significant role has been recently proposed for neuro-inflammation in the genesis of ARDS following acute brain injury. The neuro-inflammatory response represents initially a coordinated effort to protect the brain after injury, but may then become altered and be responsible for the activation of the secondary injury cascade leading to single or multiple organ dysfunction. This preclinical event may increase the susceptibility of lungs to the stress of injurious mechanical ventilation. The main targets of ventilatory management of acute brain injury patients are maintenance of an optimal oxygenation, and a tight arterial carbon dioxide control. Actual Guidelines for the management of severe traumatic brain injury, in particular, state that hypoxia (PaO2 <60 mmHg or SaO2 < 90%) should be avoided and PaCO2 level tightly controlled with a target of 35-38 mmHg. However, no published recommendation exists on which ventilator setting, in terms of tidal volume, respiratory rate, and positive end-expiratory pressure (PEEP) levels, should be used to obtain these respiratory targets. In previous studies on patients with ARDS, mechanical ventilation with a low tidal volume and moderate PEEP levels resulted in decreased mortality and increased number of ventilatory free days, and it now represents the standard of care for these patients.

Patients with acute brain injury represent a category at risk to develop ARDS both because of the adrenergic cascade and the inflammatory reaction, and because of the ventilatory strategy implemented to optimize gas exchange. Nevertheless, no clinical trial has been performed to evaluate the effect of protective ventilatory strategies upon severe acute brain injury patients.

AIMS The aim of this study is to investigate whether the application of a protective ventilatory strategy, defined as low tidal volume and moderate levels of PEEP, improves the combined end point of "event free survival" defined as survival without ventilator dependency or ARDS diagnosis, without adversely affecting neurological outcome.

Secondary aim of this study is to evaluate if protective ventilatory strategy may increase number of ventilator and organ failure free days, reduce intensive care unit (ICU) length of stay, reduce the incidence of ventilator associated pneumonia (VAP), reduce concentrations of plasma inflammatory cytokines (IL-6, TNF-alpha, TNF-RI/II, IL-8, IL-1ra, IL-1beta), without adversely affecting neurological outcome as measured by the Modified Oxford Handicap scale at intensive care unit discharge and the Glasgow Outcome Scale-extended (GOSe) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe acute brain injury (traumatic brain injury, subarachnoid haemorrhage, intra-cerebral haemorrhage, and ischemic stroke)
* Patients with not obey commands and do not open eyes on GCS (Glasgow Coma Scale)
* Less than 24 hours of mechanical ventilation (expected >72 hours)

Exclusion Criteria:

* Age < 18 years
* Diagnosis of ARDS before randomization.
* Patients unlikely to survive for the next 24 hours in the opinion of ICU consultant.
* Pregnancy
* Post-anoxic coma
* Metabolic or toxic encephalopathy
* Lack of Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of event free survival | 28 days
  Combined end point of "event free survival" defined as survival without ventilator dependency or ARDS* diagnosis
  *ARDS will be defined according to Berlin definition criteria. If chest x-ray is not immediately available, ARDS diagnosis will be suspected and confirmed later on.
  Interpretation of bilateral infiltrates on chest x-ray and of heart failure vs. fluid overload was variable and in a large observational study (LUNGSAFE, JAMA. 2016 Feb 23;315:788-800) hypoxemic patients with new infiltrates were described as a well-defined group with outcome, risk factors, comorbidities and clinical management similar to ARDS. Therefore, in March 2016 the study protocol replaced "ARDS" with "acute hypoxemic respiratory failure" as one of the components of the composite primary endpoint. Acute hypoxemic respiratory failure was defined as PaO2/FiO2 ratio < 300, with presence of infiltrates on chest x-ray, independently of lung opacities distribution and characteristics.

SECONDARY OUTCOMES:
Number of ventilator free days at 28 days | 28 days
number of ICU free days at day 28 after randomization | participants will be followed for the duration of ICU stay, an expected average of 3 weeks
Incidence of ventilator associated pneumonia (VAP) | 28 days
Cumulative SOFA free score from the randomization to day 28 | 28 days
Concentrations of plasma inflammatory cytokines | 7 days
Modify Oxford Handicap Scale at ICU discharge | participants will be followed for the duration of ICU stay, an expected average of 3 weeks
Glasgow Outcome Scale extended (GOSe) at 6 months | at 6 months
Mortality at day 28 after randomization | 28 days
LOS in ICU | 20 days (average time)
  length of stay in intensive care unit
Hospital length of stay (HLOS) | 30 days (average time)
  length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Mascia, MD, PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- University of Turin - Department of Anesthesia and Intensive care Medicine, Turin, Italy

REFERENCES:
- [Derived] Mascia L, Fanelli V, Mistretta A, Filippini M, Zanin M, Berardino M, Mazzeo AT, Caricato A, Antonelli M, Della Corte F, Grossi F, Munari M, Caravello M, Alessandri F, Cavalli I, Mezzapesa M, Silvestri L, Casartelli Liviero M, Zanatta P, Pelosi P, Citerio G, Filippini C, Rucci P, Rasulo FA, Tonetti T. Lung-Protective Mechanical Ventilation in Patients with Severe Acute Brain Injury: A Multicenter Randomized Clinical Trial (PROLABI). Am J Respir Crit Care Med. 2024 Nov 1;210(9):1123-1131. doi: 10.1164/rccm.202402-0375OC. PMID 39288368